CLINICAL TRIAL: NCT00258271
Title: A Phase I Study of CLAG Regimen in Combination With Imatinib Mesylate (Gleevec) in Refractory or Relapsed Leukemias
Brief Title: Cladribine, Cytarabine, and Imatinib Mesylate in Treating Patients With Refractory or Relapsed Acute Myeloid Leukemia or Blastic Phase Chronic Myelogenous Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000448638; URCC-U26403; URCC-RSRB-10427; NOVARTIS-CSTI571AUS161
Record Dates: First submitted 2005-11-22; First posted 2005-11-24 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia; adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult acute megakaryoblastic leukemia (M7); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia without maturation (M1); adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); blastic phase chronic myelogenous leukemia; relapsing chronic myelogenous leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Erythroblastic, Acute; Blast Crisis | interventions — Filgrastim; Cladribine; Cytarabine; Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim
Drug: cladribine
Drug: cytarabine
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cladribine and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Imatinib mesylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving cladribine and cytarabine together with imatinib mesylate may kill more cancer cells.

PURPOSE: This phase I trial is studying the side effects and best dose of imatinib mesylate when given together with cladribine and cytarabine in treating patients with refractory or relapsed acute myeloid leukemia or blastic phase chronic myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety and feasibility of cladribine, cytarabine, and imatinib mesylate in patients with refractory or relapsed acute myeloid leukemia or blastic phase chronic myelogenous leukemia.
* Determine the maximum tolerated dose of imatinib mesylate in patients treated with this regimen.
* Correlate the expression of c-kit and the presence of c-kit mutations with clinical response in patients treated with this regimen.
* Correlate the in vitro inhibitory effects of imatinib mesylate and cytarabine on the proliferation and survival of leukemic cells with clinical response in patients treated with this regimen.

OUTLINE: This is a dose-escalation study of imatinib mesylate.

Patients receive oral imatinib mesylate once daily on days 1-15 and cladribine IV over 2 hours and cytarabine IV over 4 hours on days 3-7. Patients also receive filgrastim (G-CSF) subcutaneously on days 2-7. Treatment repeats every 15 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of imatinib mesylate until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

After completion of study treatment, patients are followed periodically for up to 1 year.

PROJECTED ACCRUAL: A total of 12-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML) or blastic phase chronic myelogenous leukemia (CML)

  * Refractory AML defined as any of the following:

    * Failure to achieve complete response (CR) after 2 courses of induction chemotherapy
    * Persistent bone marrow blasts > 40% after 1 course of induction chemotherapy
    * Relapse of disease within 3 months since CR
  * Relapsed AML defined as the following:

    * Any evidence of disease recurrence after CR (early relapse occurs within 3-12 months and late relapse occurs > 12 months later)
  * No acute promyelocytic leukemia (AML-M3 FAB subgroup)

PATIENT CHARACTERISTICS:

Performance status

* ECOG 0-2

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Bilirubin ≤ 2.0 mg/dL
* AST ≤ 2.5 times upper limit of normal
* No known chronic liver disease (e.g., chronic active hepatitis or cirrhosis)

Renal

* Creatinine < 2.5 mg/dL (if 2.0-2.5 mg/dL, glomerular filtration rate must be measured and dose of cytarabine adjusted if necessary)

Cardiovascular

* No New York Heart Association grade III-IV heart disease
* No congestive heart failure
* No myocardial infarction within the past 6 months
* Ejection fraction ≥ 30%

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception during and for 3 months after completion of study treatment
* No uncontrolled systemic active infection
* No known HIV infection
* No history of allergic reaction attributed to compounds of similar chemical or biological composition to study drugs
* No history of other curatively treated malignancy except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No other concurrent biologic agents

Chemotherapy

* See Disease Characteristics
* No other concurrent chemotherapy

Endocrine therapy

* No concurrent birth control pills

Other

* More than 1 week since any prior investigational agent
* No other concurrent investigational agents or therapies
* No other concurrent anticancer agents
* No concurrent therapeutic anticoagulation with warfarin

  * Low molecular weight heparin or heparin allowed for therapeutic anticoagulation
  * Mini-dose warfarin (e.g., 1 mg per day) allowed for prophylaxis of central venous catheter thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2005-03; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille Abboud, MD, Principal Investigator — James P. Wilmot Cancer Center
Locations (1):
- James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York, United States

REFERENCES:
- [Result] Walker AR, Komrokji RS, Ifthikharuddin J, Messina P, Mulford D, Becker M, Friedberg J, Oliva J, Phillips G, Liesveld JL, Abboud C. Phase I study of cladribine, cytarabine (Ara-C), granulocyte colony stimulating factor (G-CSF) (CLAG Regimen) and simultaneous escalating doses of imatinib mesylate (Gleevec) in relapsed/refractory AML. Leuk Res. 2008 Dec;32(12):1830-6. doi: 10.1016/j.leukres.2008.04.026. Epub 2008 Jun 20. PMID 18571721